CLINICAL TRIAL: NCT02291861
Title: A Randomized, Double-Blind, Placebo-Controlled, Fixed-Dose Study of SD-809 (Deutetrabenazine) for the Treatment of Moderate to Severe Tardive Dyskinesia
Brief Title: Addressing Involuntary Movements in Tardive Dyskinesia
Acronym: AIM-TD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Auspex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SD-809-C-23; 2014-003135-19 (EudraCT Number)
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Results first posted 2018-04-11 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Tardive Dyskinesia
Keywords: Dyskinesias; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms
MeSH Terms: conditions — Tardive Dyskinesia; Dyskinesias; Movement Disorders; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms | interventions — deutetrabenazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo tablets taken twice daily for 12 weeks.
  Interventions: Drug: Placebo
- SD-809 12 mg/day (Experimental): SD-809 tablets 6 mg taken twice a day (BID) for 12 weeks.
  Interventions: Drug: SD-809
- SD-809 24 mg/day (Experimental): SD-809 tablets dose starting at 6 mg twice a day (BID) and titrated over 4 weeks to 12 mg BID. The total daily dose of 24 mg was maintained for an additional 8 weeks.
  Interventions: Drug: SD-809
- SD-809 36 mg/day (Experimental): SD-809 tablets dose starting at 6 mg twice a day (BID) and titrated over 4 weeks to 18 mg BID. The total daily dose of 36 mg was maintained for an additional 8 weeks.
  Interventions: Drug: SD-809

INTERVENTIONS:
Drug: SD-809 — SD-809 tablets dose titrated for 4 weeks until target randomized dose is reached. The dose is maintained for an additional 8 weeks. Tablets were swallowed whole with water and taken with food.
  Other Names: deutetrabenzine; Austedo
  Arms: SD-809 12 mg/day; SD-809 24 mg/day; SD-809 36 mg/day
Drug: Placebo — Placebo tablets taken twice daily for 12 weeks. Tablets were swallowed whole with water and taken with food.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether fixed-doses of an investigational drug, SD-809 (deutetrabenazine), will reduce the severity of abnormal involuntary movements of tardive dyskinesia.

ELIGIBILITY:
Inclusion Criteria:

* History of using a dopamine receptor antagonist for at least 3 months
* Clinical diagnosis of tardive dyskinesia and has had symptoms for at least 3 months prior to screening
* Subjects with underlying psychiatric diagnosis are stable and have no change in psychoactive medications
* Have a mental health provider and does not anticipate any changes to treatment regimen in the next 3 months
* History of being compliant with prescribed medications
* Able to swallow study drug whole
* Be in good general health and is expected to attend all study visits and complete study assessments
* Female subjects must not be pregnant and must agree to an acceptable method of contraception throughout the study

Exclusion Criteria:

* Currently receiving medication for the treatment of tardive dyskinesia
* Have a neurological condition other than tardive dyskinesia that may interfere with assessing the severity of dyskinesias
* Have a serious untreated or undertreated psychiatric illness
* Have recent history or presence of violent behavior
* Have unstable or serious medical illness
* Have evidence of hepatic impairment
* Have evidence of renal impairment
* Have known allergy to any component of SD-809 or tetrabenazine
* Has participated in an investigational drug or device trial and received study drug or device within 30 days
* Have acknowledged use of illicit drugs
* Have a history of alcohol or substance abuse in the previous 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2016-08-19 (Actual); Study Completion 2016-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (106):
- United States (53):
  - Teva Investigational Site 145, Tuscaloosa, Alabama
  - Teva Investigational Site 107, Anaheim, California
  - Teva Investigational Site 108, Anaheim, California
  - Teva Investigational Site 123, Glendale, California
  - Teva Investigational Site 177, Imperial, California
  - Teva Investigational Site 160, Irvine, California
  - Teva Investigational Site 106, Irvine, California
  - Teva Investigational Site 176, Loma Linda, California
  - Teva Investigational Site 121, Los Angeles, California
  - Teva Investigational Site 147, Los Angeles, California
  - Teva Investigational Site 174, Norwalk, California
  - Teva Investigational Site 170, Oceanside, California
  - Teva Investigational Site 102, Orange, California
  - Teva Investigational Site 104, San Bernardino, California
  - Teva Investigational Site 110, San Diego, California
  - Teva Investigational Site 169, San Rafael, California
  - Teva Investigational Site 129, Englewood, Colorado
  - Teva Investigational Site 139, New Haven, Connecticut
  - Teva Investigational Site 156, Washington D.C., District of Columbia
  - Teva Investigational Site 157, Boca Raton, Florida
  - Teva Investigational Site 117, Gainesville, Florida
  - Teva Investigational Site 150, Lake City, Florida
  - Teva Investigational Site 153, Miami, Florida
  - Teva Investigational Site 162, Miami, Florida
  - Teva Investigational Site 112, Orlando, Florida
  - Teva Investigational Site 144, Port Charlotte, Florida
  - Teva Investigational Site 155, Augusta, Georgia
  - Teva Investigational Site 165, Decatur, Georgia
  - Teva Investigational Site 131, Chicago, Illinois
  - Teva Investigational Site 113, Chicago, Illinois
  - Teva Investigational Site 164, Kansas City, Kansas
  - Teva Investigational Site 154, Baltimore, Maryland
  - Teva Investigational Site 101, Glen Burnie, Maryland
  - Teva Investigational Site 135, Boston, Massachusetts
  - Teva Investigational Site 118, Creve Coeur, Missouri
  - Teva Investigational Site 142, Kansas City, Missouri
  - Teva Investigational Site 175, St Louis, Missouri
  - Teva Investigational Site 161, St Louis, Missouri
  - Teva Investigational Site 178, Lincoln, Nebraska
  - Teva Investigational Site 128, Albuquerque, New Mexico
  - Teva Investigational Site 172, Commack, New York
  - Teva Investigational Site 148, New York, New York
  - Teva Investigational Site 138, Asheville, North Carolina
  - Teva Investigational Site 146, Raleigh, North Carolina
  - Teva Investigational Site 133, Charleston, South Carolina
  - Teva Investigational Site 149, Memphis, Tennessee
  - Teva Investigational Site 151, Fort Worth, Texas
  - Teva Investigational Site 115, Salt Lake City, Utah
  - Teva Investigational Site 141, Salt Lake City, Utah
  - Teva Investigational Site 168, Burlington, Vermont
  - Teva Investigational Site 171, Charlottesville, Virginia
  - Teva Investigational Site 167, Richland, Washington
  - Teva Investigational Site 166, Waukesha, Wisconsin
- Czechia (10):
  - Teva Investigational Site 559, Havířov
  - Teva Investigational Site 556, Hostivice
  - Teva Investigational Site 558, Hradec Králové
  - Teva Investigational Site 535, Litoměřice
  - Teva Investigational Site 557, Pilsen
  - Teva Investigational Site 533, Prague
  - Teva Investigational Site 532, Prague
  - Teva Investigational Site 530, Prague
  - Teva Investigational Site 531, Prague
  - Teva Investigational Site 534, Prague
- Germany (6):
  - Teva Investigational Site 502, Gera
  - Teva Investigational Site 503, Haag in Oberbayern
  - Teva Investigational Site 504, Mainz
  - Teva Investigational Site 507, Prien am Chiemsee
  - Teva Investigational Site 544, Taufkirchen
  - Teva Investigational Site 501, Wolfach
- Hungary (9):
  - Teva Investigational Site 540, Balassagyarmat
  - Teva Investigational Site 538, Budapest
  - Teva Investigational Site 541, Budapest
  - Teva Investigational Site 537, Budapest
  - Teva Investigational Site 542, Budapest
  - Teva Investigational Site 539, Doba
  - Teva Investigational Site 546, Győr
  - Teva Investigational Site 545, Kalocsa
  - Teva Investigational Site 547, Szeged
- Poland (23):
  - Teva Investigational Site 514, Bełchatów
  - Teva Investigational Site 554, Bialystok
  - Teva Investigational Site 510, Bydgoszcz
  - Teva Investigational Site 519, Bydgoszcz
  - Teva Investigational Site 536, Bydgoszcz
  - Teva Investigational Site 523, Chełmno
  - Teva Investigational Site 517, Choroszcz
  - Teva Investigational Site 513, Gdansk
  - Teva Investigational Site 512, Katowice
  - Teva Investigational Site 552, Katowice
  - Teva Investigational Site 520, Krakow
  - Teva Investigational Site 509, Krakow
  - Teva Investigational Site 508, Lodz
  - Teva Investigational Site 511, Lublin
  - Teva Investigational Site 515, Lublin
  - Teva Investigational Site 524, Lublin
  - Teva Investigational Site 549, Olsztyn
  - Teva Investigational Site 521, Pruszków
  - Teva Investigational Site 518, Sosnowiec
  - Teva Investigational Site 522, Torun
  - Teva Investigational Site 550, Warsaw
  - Teva Investigational Site 555, Warsaw
  - Teva Investigational Site 516, Wroclaw
- Slovakia (5):
  - Teva Investigational Site 529, Bratislava
  - Teva Investigational Site 525, Domaša
  - Teva Investigational Site 527, Košice
  - Teva Investigational Site 528, Rimavská Sobota
  - Teva Investigational Site 526, Rožňava

REFERENCES:
- [Result] Anderson KE, Stamler D, Davis MD, Factor SA, Hauser RA, Isojarvi J, Jarskog LF, Jimenez-Shahed J, Kumar R, McEvoy JP, Ochudlo S, Ondo WG, Fernandez HH. Deutetrabenazine for treatment of involuntary movements in patients with tardive dyskinesia (AIM-TD): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Psychiatry. 2017 Aug;4(8):595-604. doi: 10.1016/S2215-0366(17)30236-5. Epub 2017 Jun 28. PMID 28668671
- [Derived] Frank S, Anderson KE, Fernandez HH, Hauser RA, Claassen DO, Stamler D, Factor SA, Jimenez-Shahed J, Barkay H, Wilhelm A, Alexander JK, Chaijale N, Barash S, Savola JM, Gordon MF, Chen M. Safety of Deutetrabenazine for the Treatment of Tardive Dyskinesia and Chorea Associated with Huntington Disease. Neurol Ther. 2024 Jun;13(3):655-675. doi: 10.1007/s40120-024-00600-1. Epub 2024 Apr 1. PMID 38557959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at 75 study centers (38 in the US, 19 in Poland, 7 in Hungary, 6 in the Czech Republic, 3 in Slovakia, and 2 in Germany) by 75 investigators; 298 patients were enrolled.
Pre-assignment Details: Participants were randomly assigned in a 1:1:1:1 ratio to receive 1 of 3 fixed-dose regimens of SD-809 (deutetrabenazine) or placebo following a screening period.
Period: Overall Study
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
Started | 74 | 75 | 74 | 75
Safety Population | 72 | 74 | 73 | 74
Modified Intent to Treat Pop (mITT) | 58 | 60 | 49 | 55
Completed | 67 | 67 | 65 | 65
Not Completed | 7 | 8 | 9 | 10
Not completed — Adverse Event | 2 | 4 | 1 | 2
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 4
Not completed — Noncompliance | 1 | 1 | 2 | 1
Not completed — Lost to Follow-up | 2 | 1 | 4 | 0
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population was a subset of randomized participants and included all patients who were administered study drug (N=293).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day | Total
Number analyzed (Participants) | 72 | 74 | 73 | 74 | 293
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.06) | 57.0 (9.95) | 55.6 (11.34) | 58.3 (11.55) | 56.4 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 42 | 41 | 42 | 162
  Male | 35 | 32 | 32 | 32 | 131
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2 | 4
  Asian | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 15 | 19 | 10 | 56
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 59 | 58 | 54 | 61 | 232
  Other | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or latino | 7 | 6 | 3 | 7 | 23
  Not hispanic or latino | 64 | 64 | 69 | 65 | 262
  Not reported | 0 | 3 | 1 | 1 | 5
  Unknown | 1 | 1 | 0 | 1 | 3
Weight [Mean (Standard Deviation); unit: kg] | 82.8 (18.51) | 80.8 (21.00) | 86.8 (18.79) | 78.5 (17.56) | 82.2 (19.16)
Height [Mean (Standard Deviation); unit: cm] | 168.3 (9.25) | 167.7 (10.68) | 168.7 (9.39) | 167.6 (10.55) | 168.1 (9.96)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.18 (6.128) | 28.69 (6.814) | 30.64 (7.021) | 27.99 (6.178) | 29.12 (6.587)
Education Level [Count of Participants; unit: Participants]
  <= 12 years | 40 | 44 | 44 | 39 | 167
  > 12 years | 32 | 30 | 29 | 35 | 126
Time Since Tardive Dyskinesia (TD) Diagnosis [Mean (Standard Deviation); unit: years] | 6.03 (5.353) | 5.49 (5.426) | 4.98 (6.034) | 5.89 (5.342) | 5.60 (5.532)
Total Motor Abnormal Involuntary Movement Scale (AIMS) Score [Mean (Standard Deviation); unit: units on a scale] — The AIMS is an assessment tool used to detect and follow the severity of TD over time. The AIMS is composed of 12 clinician-administered and scored items.
  Total Motor assessment sums items 1 through 7 which cover orofacial movements, as well as extremity and truncal dyskinesia. Ratings were based on a 5-point scale of severity from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), to 4 (severe) for a total scale of 0-28.
  units on a scale | 8.5 (3.28) | 8.6 (3.13) | 7.7 (3.51) | 8.6 (3.84) | 8.4 (3.46)
Modified Craniocervical Dystonia Questionnaire (mCDQ-24) [Mean (Standard Deviation); unit: units on a scale] — The CDQ-24 is a disease-specific quality of life questionnaire developed for use in patients with craniocervical dystonia, including both cervical dystonia (CD) and blepharospasm (BPS). The CDQ 24 was modified such that the questions focus more directly on the impact of TD (as opposed to CD/BPS) on quality of life. Each of the 24 questions was rated by patients on a scale of 0=no impairment to 4=severest impairment for a total scale of 0 - 96. Population: One participant in the SD-809 12 mg/day group was missing a baseline mCDQ-24 total score.
  units on a scale
    number analyzed (Participants) | 72 | 73 | 73 | 74 | 292
    (all) | 40.5 (19.88) | 37.2 (20.15) | 34.4 (19.59) | 34.9 (18.34) | 36.7 (19.55)
Baseline Use of a Dopamine Receptor Antagonist (DRA) [Count of Participants; unit: Participants] — The randomization was stratified by baseline use of DRA (currently taking versus not currently taking a DRA).
  Participants
    Yes | 56 | 56 | 57 | 53 | 222
    No | 16 | 18 | 16 | 21 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Motor Abnormal Involuntary Movement Scale (AIMS) Score From Baseline to Week 12 Using a Mixed Model For Repeated Measures (MMRM)
Description: AIMS is an assessment tool used to detect and follow the severity of tardive dyskinesia (TD) over time. AIMS is composed of 12 clinician-administered and scored items. The exam was digitally video recorded using a standard protocol, and independently reviewed by blinded central raters who were experts in movement disorders.
  This outcome sums items 1 through 7 which cover orofacial movements, as well as extremity and truncal dyskinesia (the total motor AIMS score). Ratings were based on a 5-point scale of severity from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), to 4 (severe) for a total scale of 0-28. A negative change from baseline score indicates improvement.
  MMRM with treatment group, visit, treatment group-by-visit interaction, and baseline use of dopamine receptor antagonist (DRAs) as fixed effects and the baseline value as a covariate. The model was fit using an unstructured covariance structure.
Time Frame: Day 0 (Baseline), Weeks 2, 4, 8 and 12
Population: The mITT Population (N=222) included all patients in the ITT Population with a baseline AIMS score ≥6 as assessed by central video rating, were randomized to treatment, received study drug, and had at least 1 postbaseline AIMS assessment. For this outcome, participants with baseline readings and during-study readings through Week 12 are included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
Number analyzed (Participants) | 56 | 53 | 45 | 52
units on a scale | -1.4 (0.41) | -2.1 (0.42) | -3.2 (0.45) | -3.3 (0.42)
Statistical Analysis 1: Comparison: Placebo vs SD-809 36 mg/Day; A hierarchical (fixed-sequence) testing approach was used for the analysis of the primary and key secondary endpoints to maintain the experiment-wise type I error rate of 5%. The primary endpoint compared the change in total motor AIMS score from baseline to week 12 between the SD-809 36 mg/day group and the placebo group; Test type: Superiority; p = 0.001, mixed model for repeated measures — Treatment group, visit, treatment group-by-visit interaction, and baseline use of DRAs as fixed effects and the baseline value as a covariate. The model was fit using an unstructured covariance structure; LSM difference = -1.9, 95% CI 2-sided [-3.09 to -0.79] — SD-809 - placebo
Statistical Analysis 2: Comparison: Placebo vs SD-809 24 mg/Day; A hierarchical (fixed-sequence) testing approach was used for the analysis of the primary and key secondary endpoints to maintain the experiment-wise type I error rate of 5%. This key secondary endpoint compared the change in total motor AIMS score from baseline to week 12 between the SD-809 24 mg/day group and the placebo group, and is the third analysis in the fixed-sequence; Test type: Superiority; p = 0.003, mixed model for repeated measures — [p-value comment as in outcome 1, analysis 1]; LSM difference = -1.8, 95% CI 2-sided [-3.00 to -0.63] — SD-809 - placebo
Statistical Analysis 3: Comparison: Placebo vs SD-809 12 mg/Day; A hierarchical (fixed-sequence) testing approach was used for the analysis of the primary and key secondary endpoints to maintain the experiment-wise type I error rate of 5%. This key secondary endpoint compared the change in total motor AIMS score from baseline to week 12 between the SD-809 12 mg/day group and the placebo group, and is the fifth analysis in the fixed-sequence; Test type: Superiority; p = 0.217, mixed model for repeated measures — [p-value comment as in outcome 1, analysis 1]; LSM difference = -0.7, 95% CI 2-sided [-1.84 to 0.42] — SD-809 - placebo

2. Secondary Outcome: Percentage of Patients Considered a Treatment Success at Week 12 as Assessed by the Clinical Global Impression of Change (CGIC)
Description: The CGIC is a single-item questionnaire that asks the investigator to assess a patient's TD symptoms at specific visits after initiating therapy. The CGIC uses a 7 point Likert Scale, ranging from very much worse (-3) to very much improved (+3), to assess overall response to therapy.
  A treatment success was defined as "much improved" or "very much improved" at the week 12 visit.
  Patients whose status at week 12 was not known, as well as patients who were not "much improved" or "very much improved" at the week 12 visit, were considered treatment failures.
  The success 95% confidence interval (CI) was calculated with the Wilson (score) confidence limits.
Time Frame: Week 12
Population: The mITT Population (N=222) included all patients in the ITT Population with a baseline AIMS score ≥6 as assessed by central video rating, were randomized to treatment, received study drug, and had at least 1 postbaseline AIMS assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
Number analyzed (Participants) | 58 | 60 | 49 | 55
percentage of participants | 26 [16.3 to 38.4] | 28 [18.5 to 40.8] | 49 [35.6 to 62.5] | 44 [31.4 to 56.7]
Statistical Analysis 1: Comparison: Placebo vs SD-809 36 mg/Day; A hierarchical (fixed-sequence) testing approach was used for the analysis of the primary and key secondary endpoints to maintain the experiment-wise type I error rate of 5%. This key secondary endpoint compared the percentage of patients considered a treatment success at week 12 between the SD-809 36 mg/day group and the placebo group, and is the second analysis in the fixed-sequence; Test type: Superiority; p = 0.059, Cochran-Mantel-Haenszel; The statistical test was a Cochran-Mantel-Haenszel (CMH) test stratified by baseline use of dopamine receptor antagonist (DRAs); Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.960 to 4.645] — SD-809/placebo The odds ratio was the Mantel-Haenszel estimate of the common odds ratio
Statistical Analysis 2: Comparison: Placebo vs SD-809 24 mg/Day; A hierarchical (fixed-sequence) testing approach was used for the analysis of the primary and key secondary endpoints to maintain the experiment-wise type I error rate of 5%. This key secondary endpoint compared the percentage of patients considered a treatment success at week 12 between the SD-809 24 mg/day group and the placebo group, and is the fourth analysis in the fixed-sequence; Test type: Superiority; p = 0.014, Cochran-Mantel-Haenszel; The statistical test was a CMH test stratified by baseline use of DRAs; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.211 to 6.052] — SD-809/placebo The odds ratio was the Mantel-Haenszel estimate of the common odds ratio
Statistical Analysis 3: Comparison: Placebo vs SD-809 12 mg/Day; A hierarchical (fixed-sequence) testing approach was used for the analysis of the primary and key secondary endpoints to maintain the experiment-wise type I error rate of 5%. This key secondary endpoint compared the percentage of patients considered a treatment success at week 12 between the SD-809 12 mg/day group and the placebo group, and is the sixth (last) analysis in the fixed-sequence; Test type: Superiority; p = 0.734, Cochran-Mantel-Haenszel; The statistical test was a CMH test stratified by baseline use of DRAs; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.509 to 2.610] — SD-809/placebo The odds ratio was the Mantel-Haenszel estimate of the common odds ratio

3. Secondary Outcome: Change in the Modified Craniocervical Dystonia Questionnaire (mCDQ-24) Total Score From Baseline to Week 12
Description: The CDQ-24 is a disease-specific quality of life questionnaire developed for use in patients with craniocervical dystonia, including both cervical dystonia (CD) and blepharospasm (BPS). The CDQ 24 was modified such that the questions focus more directly on the impact of TD (as opposed to CD/BPS) on quality of life.
  The following domains are evaluated in the mCDQ-24: stigma, emotional well-being, pain, activities of daily living, and social/family life. Each of the 24 questions were rated by patients on a scale of 0=no impairment to 4=severest impairment for a total scale of 0 - 96. Negative change from baseline scores indicate improvement.
  For patients with missing data at week 12, the baseline or last available value was used as the week 12 value.
Time Frame: Day 0 (Baseline), Week 12
Population: The mITT Population (N=222) included all patients in the ITT Population with a baseline AIMS score ≥6 as assessed by central video rating, were randomized to treatment, received study drug, and had at least 1 postbaseline AIMS assessment. One SD-809 12 mg/day participant was missing a baseline mCDQ-24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
Number analyzed (Participants) | 58 | 59 | 49 | 55
units on a scale | -7.1 (2.06) | -5.8 (2.03) | -10.2 (2.21) | -10.7 (2.04)
Statistical Analysis 1: Comparison: Placebo vs SD-809 36 mg/Day; Test type: Superiority; p = 0.207, ANCOVA — 5% level of significance (2-sided); The statistical model was an ANCOVA with treatment group and baseline use of DRAs as fixed effects and the baseline value as a covariate; LSM difference = -3.6, 95% CI 2-sided [-9.18 to 2.00] — SD-809 - placebo
Statistical Analysis 2: Comparison: Placebo vs SD-809 24 mg/Day; Test type: Superiority; p = 0.281, ANCOVA — 5% level of significance (2-sided); [statistical method as in outcome 3, analysis 1]; LSM difference = -3.1, 95% CI 2-sided [-8.86 to 2.59] — SD-809 - placebo
Statistical Analysis 3: Comparison: Placebo vs SD-809 12 mg/Day; Test type: Superiority; p = 0.627, ANCOVA — 5% level of significance (2-sided); [statistical method as in outcome 3, analysis 1]; LSM difference = 1.3, 95% CI 2-sided [-4.10 to 6.79] — SD-809 - placebo

4. Secondary Outcome: Percentage of Patients Considered a Treatment Success at Week 12 as Assessed by the Patient Global Impression of Change (PGIC)
Description: The PGIC is a single-item questionnaire that asks the patient to assess their TD symptoms at specific visits after initiating therapy. The PGIC uses a 7 point Likert Scale, ranging from very much worse (-3) to very much improved (+3), to assess overall response to therapy. A treatment success was defined as "much improved" or "very much improved" at the week 12 visit.
  Patients whose status at week 12 was not known, as well as patients who were not "much improved" or "very much improved" at the week 12 visit, were considered treatment failures. The success 95% CI was calculated with the Wilson (score) confidence limits.
Time Frame: Week 12
Population: mITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
Number analyzed (Participants) | 58 | 60 | 49 | 55
percentage of participants | 31 [20.6 to 43.8] | 23 [14.4 to 35.4] | 45 [31.9 to 58.7] | 40 [28.1 to 53.2]
Statistical Analysis 1: Comparison: Placebo vs SD-809 36 mg/Day; Test type: Superiority; p = 0.296, Cochran-Mantel-Haenszel — 5% level of significance (2-sided); The statistical test was a CMH test stratified by baseline use of DRAs; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.694 to 3.285] — SD-809/placebo The odds ratio was the Mantel-Haenszel estimate of the common odds ratio
Statistical Analysis 2: Comparison: Placebo vs SD-809 24 mg/Day; Test type: Superiority; p = 0.134, Cochran-Mantel-Haenszel — 5% level of significance (2-sided); The statistical test was a CMH test stratified by baseline use of DRAs; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.826 to 3.994] — SD-809/placebo The odds ratio was the Mantel-Haenszel estimate of the common odds ratio
Statistical Analysis 3: Comparison: Placebo vs SD-809 12 mg/Day; Test type: Superiority; p = 0.372, Cochran-Mantel-Haenszel — 5% level of significance (2-sided); The statistical test was a CMH test stratified by baseline use of DRAs; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.302 to 1.563] — SD-809/placebo The odds ratio was the Mantel-Haenszel estimate of the common odds ratio

5. Secondary Outcome: Percentage of Participants Who Had a 50% or Greater Reduction in Total Motor Abnormal Involuntary Movement Scale (AIMS) From Baseline to Week 12
Description: Responders who had a 50% or greater improvement in total motor modified AIMS at Week 12 as compared to baseline were reported as a percentage of participants with an outcome at Week 12. The responder 95% CI is calculated with the Wilson (score) confidence limits.
  AIMS is an assessment tool used to detect and follow the severity of TD over time. AIMS is composed of 12 clinician-administered and scored items. The exam was digitally video recorded using a standard protocol, and independently reviewed by blinded central raters who were experts in movement disorders.
  This outcome sums items 1 through 7 which cover orofacial movements, as well as extremity and truncal dyskinesia (the total motor AIMS score). Ratings were based on a 5-point scale of severity from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), to 4 (severe) for a total scale of 0-28. A negative change from baseline score indicates improvement.
Time Frame: Day 0 (Baseline), Week 12
Population: mITT population of participants. Participants with missing Week 12 data were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
Number analyzed (Participants) | 58 | 60 | 49 | 55
percentage of participants | 12 [6.0 to 22.9] | 13 [6.9 to 24.2] | 35 [22.9 to 48.7] | 33 [21.8 to 45.9]
Statistical Analysis 1: Comparison: Placebo vs SD-809 36 mg/Day; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel — 5% level of significance (2-sided); The statistical test was a CMH test stratified by baseline use of DRAs; Odds Ratio (OR) = 3.80, 95% CI 2-sided [1.395 to 10.359] — SD-809/placebo The odds ratio was the Mantel-Haenszel estimate of the common odds ratio
Statistical Analysis 2: Comparison: Placebo vs SD-809 24 mg/Day; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel — 5% level of significance (2-sided); The statistical test was a CMH test stratified by baseline use of DRAs; Odds Ratio (OR) = 3.96, 95% CI 2-sided [1.460 to 10.716] — SD-809/placebo The odds ratio was the Mantel-Haenszel estimate of the common odds ratio
Statistical Analysis 3: Comparison: Placebo vs SD-809 12 mg/Day; Test type: Superiority; p = 0.829, Cochran-Mantel-Haenszel — 5% level of significance (2-sided); The statistical test was a CMH test stratified by baseline use of DRAs; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.383 to 3.316] — SD-809/placebo The odds ratio was the Mantel-Haenszel estimate of the common odds ratio

6. Secondary Outcome: Percent Change in Total Motor Abnormal Involuntary Movement Scale (AIMS) Score From Baseline to Week 12 Using a Mixed Model for Repeated Measures (MMRM)
Description: AIMS is an assessment tool used to detect and follow the severity of TD over time. AIMS is composed of 12 clinician-administered and scored items. The exam was digitally video recorded using a standard protocol, and independently reviewed by blinded central raters who were experts in movement disorders.
  This outcome sums items 1 through 7 which cover orofacial movements, as well as extremity and truncal dyskinesia (the total motor AIMS score). Ratings were based on a 5-point scale of severity from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), to 4 (severe) for a total scale of 0-28. A negative change from baseline score indicates improvement.
  MMRM with treatment group, visit, treatment group-by-visit interaction, and baseline use of DRAs as fixed effects and the baseline value as a covariate. The model was fit using an unstructured covariance structure.
Time Frame: Day 0 (Baseline), Weeks 2, 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of baseline
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
Number analyzed (Participants) | 56 | 53 | 45 | 52
percentage of baseline | -11.6 (4.32) | -20.0 (4.34) | -31.9 (4.73) | -33.1 (4.38)
Statistical Analysis 1: Comparison: Placebo vs SD-809 36 mg/Day; Test type: Superiority; p < 0.001, mixed model for repeated measures — 5% level of significance (2-sided). Treatment group, visit, treatment group-by-visit interaction, and baseline use of DRAs as fixed effects and the baseline value as a covariate. The model was fit using an unstructured covariance structure; Mean Difference (Final Values) = -21.5, 95% CI 2-sided [-33.44 to -9.52] — SD-809 - placebo
Statistical Analysis 2: Comparison: Placebo vs SD-809 24 mg/Day; Test type: Superiority; p = 0.001, mixed model for repeated measures — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -20.2, 95% CI 2-sided [-32.57 to -7.92] — SD-809 - placebo
Statistical Analysis 3: Comparison: Placebo vs SD-809 12 mg/Day; Test type: Superiority; p = 0.160, mixed model for repeated measures — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -8.4, 95% CI 2-sided [-20.15 to 3.34] — SD-809 - placebo

7. Secondary Outcome: Cumulative Percentage of Responders Based on Change in in Total Motor Abnormal Involuntary Movement Scale (AIMS) Score From Baseline to Week 12 Recorded in Incremental Steps of 10 Percentage Points
Description: AIMS is an assessment tool used to detect and follow the severity of TD over time, composed of 12 clinician-administered and scored items. The exam was digitally video recorded using a standard protocol, and independently reviewed by blinded central raters who were experts in movement disorders.
  This outcome sums items 1 through 7 which cover orofacial movements, as well as extremity and truncal dyskinesia (the total motor AIMS score). Ratings were based on a 5-point scale of severity from 0 (none), 1 (minimal), 2 (mild), 3 (moderate), to 4 (severe) for a total scale of 0-28. A negative change from baseline score indicates improvement.
  Participants with missing data are classified as non-responders. The responder 95% CI is calculated with the Wilson (score) confidence limits. If any of the expected cell counts are < 5, exact Clopper Pearson limits are presented.
  Data report the percentage of participants who responded to the percentage improvement indicated in each row.
Time Frame: Day 0 (Baseline), Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
Number analyzed (Participants) | 58 | 60 | 49 | 55
percentage of participants
  10% Improvement | 50 [37.5 to 62.5] | 62 [49.0 to 72.9] | 67 [53.4 to 78.8] | 71 [57.9 to 81.2]
  20% Improvement | 40 [28.1 to 52.5] | 47 [34.6 to 59.1] | 59 [45.2 to 71.8] | 60 [46.8 to 71.9]
  30% Improvement | 31 [20.6 to 43.8] | 32 [21.3 to 44.2] | 49 [35.6 to 62.5] | 49 [36.4 to 61.9]
  40% Improvement | 16 [8.4 to 26.9] | 23 [14.4 to 35.4] | 45 [31.9 to 58.7] | 40 [28.1 to 53.2]
  50% Improvement | 12 [6.0 to 22.9] | 13 [6.9 to 24.2] | 35 [22.9 to 48.7] | 33 [21.8 to 45.9]
  60% Improvement | 5 [1.8 to 14.1] | 7 [2.6 to 15.9] | 20 [11.5 to 33.6] | 18 [10.2 to 30.3]
  70% Improvement | 2 [0.0 to 9.2] | 3 [0.4 to 11.5] | 12 [4.6 to 24.8] | 16 [7.8 to 28.8]
  80% Improvement | 2 [0.0 to 9.2] | 2 [0.0 to 8.9] | 2 [0.1 to 10.9] | 13 [5.3 to 24.5]
  90% Improvement | 2 [0.0 to 9.2] | 0 [0.0 to 6.0] | 0 [0.0 to 7.3] | 5 [1.1 to 15.1]

8. Secondary Outcome: Participants With Adverse Events During the Overall Treatment Period
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator and includes possibly, probably and definitely related categories. Serious AEs (SAE) include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
Number analyzed (Participants) | 72 | 74 | 73 | 74
Participants
  Overall Treatment Period: any AE | 34 | 36 | 32 | 38
  Overall Treatment Period: SAE | 4 | 2 | 6 | 4
  Overall Treatment Period: Severe AE | 2 | 2 | 4 | 1
  Overall Treatment Period: treatment-related AE | 19 | 13 | 11 | 18
  Dose reduction because of AE | 0 | 0 | 1 | 3
  Dose suspension because of AE | 2 | 3 | 1 | 1
  Withdrawn from study because of AE | 2 | 4 | 2 | 3

ADVERSE EVENTS:
Time Frame: Day 1 to Week 12
Arm/Group | Placebo | SD-809 12 mg/Day | SD-809 24 mg/Day | SD-809 36 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/74 | 1/73 | 1/74
Serious Adverse Events (participants affected / at risk) | 4/72 | 2/74 | 6/73 | 4/74
Other Adverse Events (participants affected / at risk) | 14/72 | 9/74 | 9/73 | 10/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=72) | SD-809 12 mg/Day (N=74) | SD-809 24 mg/Day (N=73) | SD-809 36 mg/Day (N=74)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol interaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=72) | SD-809 12 mg/Day (N=74) | SD-809 24 mg/Day (N=73) | SD-809 36 mg/Day (N=74)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (4) | 5 (6)
Nausea (Gastrointestinal disorders) | 7 (8) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 5 (7) | 2 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data